CLINICAL TRIAL: NCT05339009
Title: Bio-adrenomedullin (Bio-ADM) as a Biomarker of Refilling in Chronic Hemodialysis Patient
Brief Title: Bio-ADM as a Biomarker of Refilling in Chronic Hemodialysis Patient
Acronym: REFILBIOADM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0068
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Disease 5D
Keywords: Chronic kidney disease; Extracorporeal purification; Bio-ADM; Vascular refilling rate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients receive conventional dialysis treatment at inclusion: All patients receive conventional dialysis treatment at inclusion
  Interventions: Biological: BioADM determination in plasma

INTERVENTIONS:
Biological: BioADM determination in plasma — BioADM determination in plasma

SUMMARY:
Aim of this study is to evaluate in a population of chronic kidney disease patients on dialysis (Stage 5D) the predictive value of bio-adrenomedullin (bio-ADM) level on vascular refilling rate.

ELIGIBILITY:
Inclusion criteria:

* Chronic Kidney Disease patient on dialysis (stage 5D) for more than 1 month
* Anuric patient

Exclusion criteria:

* Patient protected by law
* Patient under guardianship ou curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients issued from dialysis units (non profit dialysis centers)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between bio-ADM level and vascular refilling rate | Day 1
  The refilling rate will be assessed by the ratio of relative blood volume and UF max

SECONDARY OUTCOMES:
Bio-ADM value according to comorbidity factors | Day 1
  Bio-ADM value according to comorbidity factors (diabetes, heart failure and low-grade inflammation)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, MD PhD, Principal Investigator — University Hospital Center of Montpellier, FRANCE
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No